CLINICAL TRIAL: NCT06964997
Title: Anisocoria in the ICU (AICU Study): Diagnostic Implications and Clinical Outcomes
Brief Title: Anisocoria in the Intensive Care Unit (AICU Study)
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-02347; am25Sutter3
Record Dates: First submitted 2025-03-25; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Anisocoria
Keywords: Pupillary abnormality; Intensive care unit
MeSH Terms: conditions — Anisocoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective single-center cohort study aims to determine the prevalence of acute "new onset" pupillary abnormalities in adult intensive care unit patients, assess their clinical impact, identify the contexts leading to treatment changes, and evaluate their prognostic implications.

DETAILED DESCRIPTION:
Assessment of the pupil symmetry and reactivity to light are important parts of the neurological evaluation of critically ill patients in intensive care units (ICUs). Anisocoria, a condition where the pupils are unequal in size, can be found in up to 60% of patients with acute neurologic injuries. It may indicate serious underlying issues like traumatic brain injury, cerebrovascular accidents, brain tumors or viral encephalitis. However, anisocoria or impaired pupillary reactivity can also be caused from less severe conditions, such as drug effects (e.g., ipratropium bromide),Horner's syndrome after central venous cannulation, or intoxications with substances like anticholinergics, opioids, and cannabinoids. Despite these well-known causes, there is limited data on the prevalence and clinical consequences of anisocoria in ICU patients.

New onset of pupillary abnormalities often requires immediate neurological evaluation and neuroimaging (computed tomography (CT) or magnetic resonance imaging (MRI)), but many of these scans may not reveal clinically relevant findings and could expose patients to unnecessary risks. This is particularly concerning as benign causes of pupillary abnormalities are common, while more serious conditions can sometimes be overlooked. Current studies do not fully address when CT or MRI scans are necessary, or when they provide no significant clinical benefit.

This retrospective single-center cohort study has four primary objectives:

1. to determine the prevalence of acute "new onset" pupillary abnormalities (anisocoria and/or impaired light-reactive pupillary response) in adult ICU patients.
2. to assess the clinical impact of these abnormalities, particularly in terms of the frequency of diagnostic tests like CT or MRI scans, and ophthalmologic and neurologic consultations.
3. to identify when pathological findings lead to treatment modifications
4. to evaluate the prognostic implications of these pupillary abnormalities on patient outcomes.

The results of this study may improve the understanding of acute pupillary abnormalities in ICU patients, helping to optimize diagnostic strategies, reduce unnecessary neuroimaging, and enhance patient safety and outcome prediction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (i.e., patients ≥18 years of age)
* Reported incident of pupillary abnormality (either anisocoria or non-normal pupillary reactivity) in the intensive care unit at the University Hospital Basel between 2013-2024.

Exclusion Criteria:

* Patients younger than 18 years
* Patients with documented refusal of data use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (i.e., patients ≥18 years of age) with a reported incident of pupillary abnormality (either anisocoria or non-normal pupillary reactivity) in the intensive care unit at the University Hospital Basel between 2013-2024.
Sampling Method: Probability Sample
Enrollment: 920 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Acute prehospital management data | 2013-2024
  Data from acute prehospital management, as documented in emergency medical services (EMS) treatment protocols, is collected. The collected data elements are aggregated to describe the overall EMS response.
Duration of intensive care unit stay | 2013-2024
  The length of intensive care unit (ICU) stay is recorded.
Duration of hospital stay | 2013-2024
  The length of the total hospital stay is recorded.
Discharge destination | 2013-2024
  The destination at discharge is recorded.
Date of incident | 2013-2024
  The date when acute "new onset" pupillary abnormalities were first documented in patient records is recorded.
Characteristics of incident | 2013-2024
  Details on the pupillary abnormality as described in nurses' and physicians' progress notes (e.g. wording) to characterize the condition.
Type of incident | 2013-2024
  The type of pupillary abnormality (anisocoria, areactivity, or altered reaction to light) is recorded.
Additional features of the incident | 2013-2024
  Assessment of additional features related to incident of pupillary abnormality (shift type, time of day (daytime or nighttime), and environment). These features are aggregated to characterize the context in which the assault occurred.
Patient characteristics | 2013-2024
  Information on the patient (e.g., principal diagnosis, comorbidities, medication) is documented.
Consequences of the Incident | 2013-2024
  Evaluation of medical assessments and interventions following the incident, including Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) scans, ophthalmologic or neurologic consultations.
Comprehensive assessment of the neurological status based on validated clinical assessment | 2013-2024
  Neurological status during ICU stay is assessed using available data in the patient register from validated neurological assessments. These may include the Richmond Agitation-Sedation Scale (RASS), Sedation-Agitation Scale (SAS), Glasgow Coma Scale (GCS), Intensive Care Delirium Screening Checklist (ICDSC), or Status Epilepticus Severity Score (STESS). The specific tool used, as well as the scale of the score and meaning behind the score, depends on routine clinical practice and available documentation in the register. If multiple scores are available for a patient, they will be aggregated to provide a comprehensive assessment of neurological status. This outcome will be reported as a descriptive summary, synthesizing findings across tools, rather than as a single quantitative score.
Comprehensive assessment of critical illness severity based on standardized scoring systems | 2013-2024
  Disease severity during ICU stay is assessed using standardized scoring systems, including the Acute Physiology and Chronic Health Evaluation II (APACHE II), Simplified Acute Physiology Score II (SAPS II), and Sequential Organ Failure Assessment (SOFA), depending on data availability in the patient register. The specific scoring system applied, as well as the scale and interpretation of the score, varies based on routine clinical practice and available documentation. Where multiple severity scores are available, they will be synthesized to provide a descriptive summary of overall illness severity rather than a single quantitative score.
Charlson Comorbidity Index | 2013-2024
  The Charlson Comorbidity Index (CCI) is calculated based on pre-existing comorbidities and additional diagnoses. The CCI predicts the ten-year mortality for a patient who may have a range of comorbid conditions. It assigns weighted scores (from 0 to maximal 6) to 17 comorbid conditions (e.g., heart disease, diabetes, cancer), resulting in a total score ranging from 0 to 33, if the patient had the most severe form of each of the 17 conditions.
Laboratory parameters | 2013-2024
  Routine laboratory value for e.g. C-Reactive Protein (CRP), albumin, Lactate Dehydrogenase (LDH), Creatine Kinase (CK), procalcitonin, white blood cell levels, creatinine, liver enzymes, blood gas analyses, metabolic data, and toxicologic screenings, is collected. The specific parameters recorded may vary depending on the laboratory assessments documented in the patient register. All values will be reported using their respective units of measurement.These parameters are aggregated to support an overall clinical interpretation rather than a single numerical value. This approach reflects standard clinical practice, where multiple lab values are considered together to assess a patient's condition.
Glasgow Outcome Score | 2013-2024
  The Glasgow Outcome Score (GOS) is calculated based on the assessment of key clinical outcomes such as inhospital mortality, survival, survival with neurofunctional alteration, return to premorbid neurological function, and hospital readmission to determine the patient outcome.
  The GOS ranges from 1 (death) to 5 (good recovery).
Therapeutic intervention | 2013-2024
  The therapeutic intervention is document, including information on duration, dosage and number of treatment medication, number of neuroleptic, sedative and analgesic drugs, use of ipratropium bromide, invasive procedures, such as intubation, mechanical, ventilation, vasopressors, installation of central lines, i.v. thrombolysis, endovascular thrombectomy, surgical hemicraniectomy, insertion of ventricular drains, intracranial pressure monitoring, i.v. administration of mannitol or saline, nutrition, etc.
Vital signs | 2013-2024
  Vital signs are analyzed based on the data available in the patient register. These may include blood pressure, heart rate, respiratory rate, oxygen saturation, body temperature, level of consciousness, intracranial pressure, and drainage rate of cerebrospinal fluid. The specific parameters recorded depend on the clinical documentation available. All values will be reported using their respective units of measurement. These values are aggregated to support an overall clinical assessment rather than a single numerical score. This reflects standard practice, where multiple vital signs are interpreted together to evaluate a patient's condition.
Fluid balance data | 2013-2024
  Fluid balance data, including the administration of fluids such as blood products, crystalloids, and enteral/parenteral nutrition, are documented. These components are aggregated to represent overall fluid input for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, Prof. Dr. med., Principal Investigator — University Hospital Basel, Clinic for Intensive Care Medicine
Locations (1):
- University Hospital Basel, Clinic for Intensive Care Medicine, Basel, Canton of Basel-City, Switzerland